CLINICAL TRIAL: NCT04503018
Title: Psychological Effects of Implant Loss
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-06214
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female
Keywords: Breast reconstruction; Plastic surgery; Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Interviewed -implant loss: Patients who have had immediate breast reconstruction and lost the implant due to for example infection.
- Questionnaires - implant loss: Patients who have had immediate breast reconstruction and lost the implant due to for example infection.
- Questionnaires - controls: Patients who have had immediate breast reconstruction without complications

SUMMARY:
Previous quality of life studies have suggested that long term satisfaction with breast reconstruction may be affected by postoperative complications. Complication frequencies, especially the risk for implant loss, is considerably higher in immediate than in delayed breast reconstruction. Knowledge about how implant loss affects the patient's experience of her breast reconstruction can guide us in the choice between immediate and delayed breast reconstruction in high risk patients and help us better prepare the patients for possible complications. This study will investigate patients' experiences with losing an implant in connection with immediate breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Biological women
* Age >18 years
* Have lost an implant after a mastectomy and immediate breast reconstruction

Exclusion Criteria:

* Inability to give informed consent
* inability to speak and understand Swedish
* relapse of breast cancer after the reconstruction
* metastatic disease
* psychiatric co-morbidity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Purposive criterion sampling technique is used. The population will identified through an operation planning software
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Experiences and psychological effects of implant loss after immediate breast reconstruction | 10 years
  Interviews
Effect on quality of life of implant loss: scale | 10 years
  Breast-Q reconstruction post-operative. It includes different domains: health-related quality of life (HR-QOL; including physical, psychosocial, and sexual well-being) and patient satisfaction (including satisfaction with breasts, outcome, and care). Each scale produces an independent score from 0-100.a higher score means greater satisfaction or better QOL
Effect on body image of implant loss | 10 years
  Body-Esteem Scale for Adolescents and Adults (BESAA). It consists of three subscales: BE-appearance, BE-weight and BE-attribution.The scale has 23 items and the respondents indicated their degree of agreement on a 5-point Likert scale ranging from 0 (never) to 4 (always).High score indicates higher dimensions of the Body Esteem.
Effect on depression and anxiety of implant loss | 10 years
  Hospital Anxiety and Depression scale (HAD).The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression.For both scales, scores of less than 7 indicate non-cases. 8-10 mild, 11-14 moderate, 15-21 severe.
Coping strategies | 10 years
  Brief-cope, a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event.Scores are presented for the two overarching coping styles: avoidant and approach.The scale can determine someone's primary coping styles.
Coping strategies | 10 years
  The Life orientation test - revised (Lot-R) is a 10-item scale that measures how optimistic or pessimistic people feel about the future. High values imply optimism.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Hansson, PhD, Principal Investigator — Göteborg University
Locations (1):
- Västra Götaland, Gothenburg, Sweden

REFERENCES:
- [Result] Weick L, Ericson A, Sandman L, Bostrom P, Hansson E. Patient experience of implant loss after immediate breast reconstruction: An interpretative phenomenological analysis. Health Care Women Int. 2023 Jan;44(1):61-79. doi: 10.1080/07399332.2021.1944152. Epub 2021 Aug 24. PMID 34427538
- [Result] Weick L, Lunde C, Hansson E. The effect of implant loss after immediate breast reconstruction on patient satisfaction with outcome and quality of life after five years - a case-control study. J Plast Surg Hand Surg. 2023 Feb-Dec;57(1-6):263-270. doi: 10.1080/2000656X.2022.2061501. Epub 2022 Apr 15. PMID 35427208
- See also: Full text article — http://liu.diva-portal.org/smash/get/diva2:1591756/FULLTEXT01.pdf